CLINICAL TRIAL: NCT03641079
Title: Identification of Compound From Brinjal Peel Extract That is Effective in the Treatment of Severe Palmar Arsenical Keratosis and Bowen's Disease
Brief Title: Identification of Compound From Brinjal Peel Extract in the Treatment of Palmar Arsenical Keratosis and Bowen's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Razia Sultana, Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: No.BSMMU/2018/2961
Record Dates: First submitted 2018-08-18; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-04

CONDITIONS: Keratotic Nodular Size

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- brinjal peel extract containing cream (Experimental): intervention-brinjal peel extract containing cream, dose-twice daily for 12 weeks
  Interventions: Drug: Brinjal peel extract containing cream

INTERVENTIONS:
Drug: Brinjal peel extract containing cream — Brinjal peel extract, white wax, white petrolatum, stearyl alcohol

SUMMARY:
Arsenicosis is a major health problem in Bangladesh. Long term exposure of arsenic causes keratosis of palm which reduce working capacity of patient. It also causes invasive skin lesions like Bowen's disease which has a risk to develop squamous cell carcinoma. Brinjal peel is well known for its antioxidant and anticancer properties. So this study will be conducted to identify the compound from brinjal peel extract and to see its outcome on keratosis and Bowen's disease.

DETAILED DESCRIPTION:
Arsenicosis is a major health problem in Bangladesh. About half of the population are chronically exposed to high concentration of arsenic through contaminated drinking water. In arsenicosis, keratosis of palm and sole occur which reduce the working capacity of the patient and affect the socioeconomic condition. It also causes invasive skin lesions like Bowen's disease, squamous cell carcinoma, and basal cell carcinoma. Bowen's disease usually appears as a persistent reddened scaly patch on the skin and has a risk (3-5%) to develop squamous cell carcinoma. Keratosis can be treated by different topical preparations like salicylic acid, propylene glycol and oral antioxidant, zinc and folic acid, but treatment by these medicines require a longer time to relieve and thus reduce patient's compliance. On the other hand, treatment options available for Bowen's disease are expensive. Brinjal is a common vegetable which contains steroidal alkaloids, steroidal glycosides, delphinidine, nasunin and other biologically active compounds. These biologically active compounds are effective against human cancer cells by various mechanisms. One study shows that a topical cream prepared from brinjal peel extract is effective in keratosis and skin carcinoma. So, this study will be conducted to see the outcome of brinjal peel extract in severe palmar arsenical keratosis and Bowen's disease and to identify the compound that is responsible for the effect. The study will be an Open Phase- II Clinical Trial. It will be conducted in Bangabandhu Sheikh Mujib Medical University and Bhanga Upazilla of Faridpur District. Extracts from brinjal peel will be collected by using a mixture of ethanol, chloroform and acetic acid as a solvent in Soxhlet extractor and rotary evaporator. Thin Layer Chromatography (TLC), Nuclear Magnetic Resonance (NMR) and Infrared (IR) of extract will be done to identify compound. Cytotoxicity assay will be done by using brine shrimp bioassay. Then a topical cream will be prepared from the extract and supplied at the field level through a temporary arsenic clinic at an interval of two weeks. Instruction will be given to the patients about applying the cream. Adherence and adverse effects of the cream will be monitored regularly through phone calls and during each visit. Photograph will be taken and size of the keratotic nodules as well as, lesions of Bowen's disease will be measured before the start and after completion of treatment. Clinical improvement will be assessed by the mean scoring of nodules and lesions and perception of patients about their improvement by using Likert Scale. Statistical analysis and results will be presented in tabulated forms and in different diagrams.

ELIGIBILITY:
Inclusion Criteria:

* Presence of severe keratosis and/or Bowen's disease
* Drinking arsenic contaminated water for at least six months
* Patient voluntarily agreed to participate

Exclusion Criteria:

* Age less than 18 years or more than 60 years
* Pregnant and nursing mother
* Skin diseases like atopic dermatitis, eczema and psoriasis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-09-16 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Keratotic nodular size and lesion size of Bowen's disease | 12 weeks
  Nodular size and lesion size will be measured by slide calipers

CONTACTS AND LOCATIONS:
Overall Officials: Razia Sultana, MBBS, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Faridpur, Bhanga, Hamirdi Community Clinic, Bangladesh